CLINICAL TRIAL: NCT01790048
Title: Comparison of a Novel Ready-to-use Supplementary Food (RUSF) With Whey Permeate to Standard Peanut/Soy RUSF for the Treatment of Moderate Acute Malnutrition in Rural Malawian Children: a Randomised, Double-blinded, Clinical Effectiveness Trial
Brief Title: Whey Permeate Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201211066
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2018-07

CONDITIONS: Malnutrition
Keywords: MAM
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey permeate RUSF (Experimental): 75 kcal/kg/day (314 k Joules (kJ)/kg/day) of whey RUSF. Whey RUSF contains whey permeate, Whey Permeate (WPC) 80 (contains at least 80% protein), peanut paste, sugar, soy oil, a customized micronutrient premix to account for the minerals in whey permeate, and an emulsifier. Whey permeate RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Interventions: Dietary Supplement: Whey permeate RUSF
- Soy Protein RUSF (Active Comparator): 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. Soy RUSF contains extruded soy flour, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate (Roche, Mumbai, India). Soy RUSF has no protein from animal sources. Soy RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Interventions: Dietary Supplement: Soy Protein RUSF

INTERVENTIONS:
Dietary Supplement: Whey permeate RUSF — Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Whey RUSF contains whey permeate, WPC 80 (contains at least 80% protein), peanut paste, sugar, soy oil, a customized micronutrient premix to account for the minerals in whey permeate, and an emulsifier.
  Arms: Whey permeate RUSF
Dietary Supplement: Soy Protein RUSF — Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of soy RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Soy RUSF contains extruded soy flour, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate (Roche, Mumbai, India). Soy RUSF has no protein from animal sources.
  Arms: Soy Protein RUSF

SUMMARY:
This is a prospective, randomized, double-blinded, controlled clinical effectiveness trial of two supplementary foods in the treatment of MAM.

Specific Aim 1: Test the effectiveness of two supplementary foods, whey RUSF and soy RUSF, in the treatment of MAM in 6-59 month old children in a 12-week home-based supplementary feeding program.

Hypothesis: The proportion of children who recover receiving either soy or whey RUSF will differ by no more than three percent.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded, controlled clinical effectiveness trial assessing the treatment of moderate acute malnutrition (MAM) with one of two supplementary foods for a period of up to 12 weeks. The overall purpose of this research is to see if your child will grow and gain weight more rapidly using one of two peanut butter foods as he/she recovers from protein-energy malnutrition.

Subjects will be given a soy or dairy peanut butter food at their home. The peanut butter food has either small amounts of soya protein and minerals (iron, zinc) or whey powder and minerals added to them. Subjects will have enough food to feed the child for 2 weeks, and asked to return every 2 weeks to be weighed, measured and given more food. The parents of the subjects will be asked to feed their child this food until his/her weight has returned to what is considered normal for the child's height. Subjects will then return after 3, 6 and 12 months for a check-up. At these check-ups, he/she will be measured and examined.

The current standard of care is to allow the child to recover without food or with supplemental flour thus all participation is related to research. Participation in this study is expected to last 8-12 weeks of therapy with follow up in 12 months after completion of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children with MAM defined as mid-upper-arm circumference, MUAC, ≤ 12.5 cm and > 11.5 cm without bipedal edema.

Exclusion Criteria:

* Children simultaneously involved in another research trial or supplemental feeding program
* Children with developmentally delayed
* Children with a chronic debilitating illness such as cerebral palsy (not including HIV or TB)
* Children with a history of peanut or milk allergy
* Children will also be excluded if they had received therapy for acute malnutrition within one month prior to presentation.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2259 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Project Peanut Butter, Blantyre, Malawi

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Caulfield LE, de Onis M, Blossner M, Black RE. Undernutrition as an underlying cause of child deaths associated with diarrhea, pneumonia, malaria, and measles. Am J Clin Nutr. 2004 Jul;80(1):193-8. doi: 10.1093/ajcn/80.1.193. PMID 15213048
- [Background] Shankar AH. Nutritional modulation of malaria morbidity and mortality. J Infect Dis. 2000 Sep;182 Suppl 1:S37-53. doi: 10.1086/315906. PMID 10944483
- [Background] Ezzati M, Lopez AD, Rodgers A, Vander Hoorn S, Murray CJ; Comparative Risk Assessment Collaborating Group. Selected major risk factors and global and regional burden of disease. Lancet. 2002 Nov 2;360(9343):1347-60. doi: 10.1016/S0140-6736(02)11403-6. PMID 12423980
- [Background] George E, Noel F, Bois G, Cassagnol R, Estavien L, Rouzier Pde M, Verdier RI, Johnson WD, Pape JW, Fitzgerald DW, Wright PF. Antiretroviral therapy for HIV-1-infected children in Haiti. J Infect Dis. 2007 May 15;195(10):1411-8. doi: 10.1086/514823. Epub 2007 Apr 3. PMID 17436220
- [Background] Matilsky DK, Maleta K, Castleman T, Manary MJ. Supplementary feeding with fortified spreads results in higher recovery rates than with a corn/soy blend in moderately wasted children. J Nutr. 2009 Apr;139(4):773-8. doi: 10.3945/jn.108.104018. Epub 2009 Feb 18. PMID 19225128
- [Background] Nackers F, Broillet F, Oumarou D, Djibo A, Gaboulaud V, Guerin PJ, Rusch B, Grais RF, Captier V. Effectiveness of ready-to-use therapeutic food compared to a corn/soy-blend-based pre-mix for the treatment of childhood moderate acute malnutrition in Niger. J Trop Pediatr. 2010 Dec;56(6):407-13. doi: 10.1093/tropej/fmq019. Epub 2010 Mar 23. PMID 20332221
- [Background] Lagrone L, Cole S, Schondelmeyer A, Maleta K, Manary MJ. Locally produced ready-to-use supplementary food is an effective treatment of moderate acute malnutrition in an operational setting. Ann Trop Paediatr. 2010;30(2):103-8. doi: 10.1179/146532810X12703901870651. PMID 20522296
- [Background] LaGrone LN, Trehan I, Meuli GJ, Wang RJ, Thakwalakwa C, Maleta K, Manary MJ. A novel fortified blended flour, corn-soy blend "plus-plus," is not inferior to lipid-based ready-to-use supplementary foods for the treatment of moderate acute malnutrition in Malawian children. Am J Clin Nutr. 2012 Jan;95(1):212-9. doi: 10.3945/ajcn.111.022525. Epub 2011 Dec 14. PMID 22170366
- [Background] Myatt M, Khara T, Collins S. A review of methods to detect cases of severely malnourished children in the community for their admission into community-based therapeutic care programs. Food Nutr Bull. 2006 Sep;27(3 Suppl):S7-23. doi: 10.1177/15648265060273S302. PMID 17076211
- [Background] Knueppel D, Demment M, Kaiser L. Validation of the Household Food Insecurity Access Scale in rural Tanzania. Public Health Nutr. 2010 Mar;13(3):360-7. doi: 10.1017/S1368980009991121. Epub 2009 Aug 26. PMID 19706211
- [Background] Manary MJ. Local production and provision of ready-to-use therapeutic food (RUTF) spread for the treatment of severe childhood malnutrition. Food Nutr Bull. 2006 Sep;27(3 Suppl):S83-9. doi: 10.1177/15648265060273S305. PMID 17076214
- [Result] Stobaugh HC, Ryan KN, Kennedy JA, Grise JB, Crocker AH, Thakwalakwa C, Litkowski PE, Maleta KM, Manary MJ, Trehan I. Including whey protein and whey permeate in ready-to-use supplementary food improves recovery rates in children with moderate acute malnutrition: a randomized, double-blind clinical trial. Am J Clin Nutr. 2016 Mar;103(3):926-33. doi: 10.3945/ajcn.115.124636. Epub 2016 Feb 10. PMID 26864368

RESULTS

PARTICIPANT FLOW:
Groups:
- Whey Permeate RUSF: 75 kcal/kg/day (314 k Joules (kJ)/kg/day) of whey RUSF. Whey RUSF contains whey permeate, Whey Permeate (WPC) 80 (contains at least 80% protein), peanut paste, sugar, soy oil, a customized micronutrient premix to account for the minerals in whey permeate, and an emulsifier. Whey permeate RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Whey permeate RUSF: Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Whey RUSF contains whey permeate, WPC 80 (contains
- Soy Protein RUSF: 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. Soy RUSF contains extruded soy flour, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate (Roche, Mumbai, India). Soy RUSF has no protein from animal sources. Soy RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Soy Protein RUSF: Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of soy RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Soy RUSF contains extruded soy
Period: Overall Study
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Started | 1156 | 1103
Completed | 1144 | 1086
Not Completed | 12 | 17
Not completed — Incorrect Age | 9 | 14
Not completed — data entry error | 0 | 1
Not completed — Other | 0 | 2
Not completed — SAM at Enrollment | 2 | 0
Not completed — Measurement error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF | Total
Number analyzed (Participants) | 1144 | 1086 | 2230
Age, Continuous [Median (Standard Deviation); unit: months] | 16.4 (9.3) | 16.5 (8.9) | 16.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 688 | 639 | 1327
  Male | 456 | 447 | 903
MUAC, cm [Median (Standard Deviation); unit: cm] | 12.1 (.27) | 12.1 (.27) | 12.1 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Recovery From Moderate Acute Malnutrition (MAM)
Description: The primary outcome measures will be recovery from MAM (achieving MUAC ≥ 12.5 cm by 12 weeks) or failure (death, development of severe acute malnutrition, transfer to hospital for inpatient care, failure to recover from MAM by 12 weeks, default).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
Participants | 960 | 874

2. Secondary Outcome: Weight
Description: Amount of weight gained over the course of treatment
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Gain (g/kg/day)
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
Gain (g/kg/day) | 2.95 (2.04) | 2.79 (2.16)

3. Secondary Outcome: Height
Description: Amount of height gained over the intervention period.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm/d
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
mm/d | 0.30 (0.28) | 0.29 (0.29)

4. Secondary Outcome: Mid-Upper-Arm Circumference (MUAC) Gain
Description: Gain in mid-upper arm circumference
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm/d
Groups:
- Whey Permeate RUSF: 75 kcal/kg/day (314 k Joules (kJ)/kg/day) of whey RUSF. Whey RUSF contains whey permeate, Whey Permeate (WPC) 80 (contains at least 80% protein), peanut paste, sugar, soy oil, a customized micronutrient premix to account for the minerals in whey permeate, and an emulsifier. Whey permeate RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.Whey permeate RUSF: Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Whey RUSF contains whey permeate, WPC 80 (contains at
- Soy Protein RUSF: 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. Soy RUSF contains extruded soy flour, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate (Roche, Mumbai, India). Soy RUSF has no protein from animal sources. Soy RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Soy Protein RUSF: Each child will receive 75 kcal/kg/day (314kJ/kg/day) of soy RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Soy RUSF contains extruded soy flo
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
mm/d | 0.26 (0.27) | 0.22 (0.28)

5. Secondary Outcome: Time to Graduation
Description: The amount of time required for a patient to reach recovery
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
days | 29.3 (19.0) | 30.4 (20.1)

6. Secondary Outcome: Adverse Events
Description: Any adverse events from the supplementary foods reported in the 3 month time frame.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Number analyzed (Participants) | 1144 | 1086
Participants | 0 | 0

ADVERSE EVENTS:
Groups:
- Soy Protein RUSF: 75 kcal/kg/day (314 kJ/kg/day) of whey RUSF. Soy RUSF contains extruded soy flour, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate (Roche, Mumbai, India). Soy RUSF has no protein from animal sources. Soy RUSF will be locally produced and will undergo quality assurance and safety testing for aflatoxin and microbial contamination at the Malawi Bureau of Standards and Eurofins Scientific Inc., Des Moines, Iowa, USA.
  Soy Protein RUSF: Each child will receive 75 kcal/kg/day (314 kJ/kg/day) of soy RUSF. A ration of sufficient for two weeks based on the subject's weight will be distributed at each visit. Children will be asked to return every two weeks for follow-up, where caretakers report on the child's clinical symptoms, anthropometric measurements are re-assessed, and additional supplementary food is distributed for those that remained wasted.
  Soy RUSF contains extruded soy f
Arm/Group | Whey Permeate RUSF | Soy Protein RUSF
Serious Adverse Events (participants affected / at risk) | 0/1144 | 0/1086
Other Adverse Events (participants affected / at risk) | 0/1144 | 0/1086

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes